CLINICAL TRIAL: NCT04144153
Title: Opioid Free Total Intravenous Anesthesia Within an Enhanced Recovery After Surgery Pathway for Bariatric Surgery: A Randomized Controlled Clinical Trial
Brief Title: Opioid Free Anesthesia and Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 19-0728
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Quality of Recovery
MeSH Terms: interventions — Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Free Anesthesia Group (Experimental)
  Interventions: Combination Product: Opioid Free Total Intravenous Anesthesia
- Opioid Anesthesia Group (Active Comparator)
  Interventions: Combination Product: Total Intravenous anesthesia with opioid

INTERVENTIONS:
Combination Product: Opioid Free Total Intravenous Anesthesia — Total intravenous anesthesia with propofol and dexmedetomidine hydrochloride and ketamine hydrochloride
  Arms: Opioid Free Anesthesia Group
Combination Product: Total Intravenous anesthesia with opioid — Total Intravenous anesthesia with opioid
  Arms: Opioid Anesthesia Group

SUMMARY:
The morbidly obese bariatric surgery population is susceptible to opioid-induced complications such as respiratory depression and postoperative nausea and vomiting. This population may in particular benefit from opioid-sparing or opioid-free anesthetic techniques. This study aims to evaluate the effect of opioid free total intravenous anesthesia on postoperative quality of recovery in patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Non-pregnant
* Undergoing laparoscopic bariatric surgery for weight loss.

Exclusion Criteria:

* Unable to obtain informed consent or consent withdrawn.
* Patients who are pregnant or nursing.
* ASA IV-V
* Alcohol or narcotic misuse or dependence in the last 2 years.
* Preoperative daily opioid use for one year for pain management.
* Egg or soy product allergy
* Active liver disease
* Patients with left ventricular assist devices
* Abnormal renal function
* Any contraindication to any opioid or non-opioid pain analgesics
* Any physical, mental or medical condition that in the opinion of the investigator, makes study participation inadvisable.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery | Up to two postoperative weeks
  Quality of Recovery (QoR-15), a patient-reported outcome questionnaire that assesses the quality of functional recovery after surgery and anesthesia with a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery).

SECONDARY OUTCOMES:
Pain Intensities | Up to postoperative day one
  Postoperative pain intensities using a 0 to 10 numerical rating scale (NRS) with higher scores indicative of higher pain intensities.
Opioid Consumption | Up to postoperative day one
  Total postoperative opioid consumption
Time to Aldrete Score of 9 | Up to postoperative day one
  Time to post-anesthesia care unit discharge readiness

OTHER OUTCOMES:
Postoperative Nausea and Vomiting | Up to postoperative day one
  The incidence of any postoperative nausea, retching, or vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Aronsohn, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No